CLINICAL TRIAL: NCT00106756
Title: Familial Exudative Vitreoretinopathy Clinical and Molecular Studies
Brief Title: Clinical and Genetic Studies of Familial Exudative Vitreoretinopathy
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050104; 05-EI-0104
Record Dates: First submitted 2005-03-29; First posted 2005-03-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-06-26

CONDITIONS: Exudatiaon; Avascular Retina; Retina Fold; Eye Diseases; Familial Exudative Vitreoretinopathy; FEVR
Keywords: Exudation; Avascular Retina; Retina Fold
MeSH Terms: conditions — Eye Diseases; Familial Exudative Vitreoretinopathies

SUMMARY:
This study will examine the extent of the vision problem in familial exudative vitreoretinopathy (FEVR) and try to identify the genes responsible for this hereditary eye disorder. Patients with FEVR have incomplete formation of blood vessels in the periphery of the retina (the inner part of the eye that is responsible for vision). As a result, abnormal vessels can form and retinal detachment and vitreous bleeding can occur, causing significant vision loss. Vision loss usually begins in childhood, gradually worsening over time. Some patients eventually become blind.

Patients of all ages with FEVR and their family members may be eligible for this study. Participants undergo the following tests and procedures:

* Family history, especially regarding eye disease. A family tree is drawn.
* Blood draw for genetic testing related to FEVR.
* Eye examination to assess visual acuity (eye chart test) and eye pressure, and to examine pupils, lens, retina and eye movements. The pupils are dilated with drops for this examination.
* Fluorescein angiography to evaluate the eye's blood vessels. A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina are taken using a camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible blood vessel abnormality.
* Patients affected with FEVR will also undergo DEXA scan to look for osteoporosis. X-rays are used to scan the hip, forearm and spine for bone density measurements.

DETAILED DESCRIPTION:
Background: Familial exudative vitreoretinopathy (FEVR) is a rare hereditary disorder of the retinal vasculature characterized by abrupt cessation of the growth of peripheral retinal capillaries. FEVR seems to exhibit significant phenotypic and genotypic variability but since this is a rare disease the clinical and genetic characteristics of the disease have not been extensively studied so far. Correlation of phenotypes with certain genotypes have not been made yet. Clinical findings can vary from very mild disease with only subtle changes of the peripheral retinal vasculature without symptoms to severe disease with retinal neovascularization, retinal exudates, vitreoretinal adhesions, peripheral vitreous opacities, retinal folds and tractional retinal detachment. The condition remarkably resembles retinopathy of prematurity but affected patients do not have a history of prematurity or supplementary oxygen use.

The disorder is usually inherited as an autosomal dominant trait but few families show x-linked or autosomal recessive inheritance. A significant number of patients with autosomal dominant FEVR show linkage to 11q13-q23 (EVR1). Two genes in this locus have recently been shown to be associated with the disease. FZD4, the gene that encodes for Frizzled-4, the Wnt receptor, is one of them. It has been estimated by recent studies that 20-30% of patients with autosomal dominant FEVR show mutations in FZD4. LRP5 (low-density-lipoprotein receptor-related protein 5), a Wnt co-receptor, was recently shown to be mutated in approximately 15% of cases. One large autosomal dominant pedigree has shown linkage to 11p13-p12 locus (EVR3) and this gene has not yet been identified. It now becomes obvious that more genes are associated with the autosomal dominant type of the disease. Most of the patients with the x-linked type have mutations in the Norrie disease gene (EVR2). The autosomal recessive form of the disease is much rarer and linkage studies have not yet been performed.

Aims: The objectives of this protocol are to study the clinical characteristics of FEVR, and also to assist in identifying the location and sequence of corresponding genes. Since one of the genes so far identified, LRP5, is also causing the osteoporosis-pseudoglioma syndrome, an inherited disorder with severe osteoporosis, we would also like to know if FEVR patients, especially those with mutations in LRP5 also have some degree of osteoporosis. Localization and identification of the responsible gene will help us understand the pathogenesis of FEVR and possibly the mechanism of retinal angiogenesis and lead to potential treatments.

Methods: Patients as well as available family members are to be evaluated by physical examination and fluorescein angiography, in order to clinically characterize the inheritance pattern in each family. Blood will be obtained by all participating subjects for the molecular studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

The patients must carry the clinical diagnosis of familial exudative vitreoretinopathy. Whenever a patient fulfills the above requirement additional family members can be included in the study as participants. Subjects of any ethnic background, gender, age, sexual orientation, or health status will be included.

EXCLUSION CRITERIA:

Prematurity and supplemental oxygen use at bith can cause a clinical picture similar to familial exudative vitreoretinopathy. The existence of either of those factors in the past medical history of a patient will necessitate exclusion from the study. Since fluorescein angiography is crucial for the correct diagnosis of the syndrome, patients with a previous allergic reaction to fluorescein dye will also be excluded. Patients inability or unwillingness to provide a blood sample is an exclusion criterion as well.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105
Dates: Start 2005-03-18; Primary Completion 2006-11-01 (Actual); Study Completion 2006-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Izaak Walton Killam Grace Health Centre, Halifax, Canada
- St. James University, Leeds, United Kingdom

REFERENCES:
- [Background] Criswick VG, Schepens CL. Familial exudative vitreoretinopathy. Am J Ophthalmol. 1969 Oct;68(4):578-94. doi: 10.1016/0002-9394(69)91237-9. No abstract available. PMID 5394449
- [Background] Gow J, Oliver GL. Familial exudative vitreoretinopathy. An expanded view. Arch Ophthalmol. 1971 Aug;86(2):150-5. doi: 10.1001/archopht.1971.01000010152007. No abstract available. PMID 5571414
- [Background] Laqua H. Familial exudative vitreoretinopathy. Albrecht Von Graefes Arch Klin Exp Ophthalmol. 1980;213(2):121-33. doi: 10.1007/BF00413539. PMID 6906151